Date: 2<sup>nd</sup> August 2022

Comparison of preoperative analgesics on the efficacy of inferior alveolar nerve block on patients with symptomatic irreversible pulpitis: a double blinded, randomized controlled trial.

## **Statistical Analysis Plan:**

Test of normality was checked using one sample Shapiro Wilk. One-way ANOVA with Tukey's post-hoc will be employed if parametric test criteria is met; however, if the parametric criteria was not fulfilled, the experimental groups will be compared using Kruskal–Wallis test with post-hoc analysis. The Chi-square test will be used to compare gender and drug groups against the IANB efficacy. These aforementioned tests were conducted on SPSS Statistics version 25 (IBM Corp., Armonk, NY, USA).